CLINICAL TRIAL: NCT02423018
Title: Evaluation of Pregabalin's Abuse Liability and Its Effects on Benzodiazepine Withdrawal Symptoms in Inpatients Undergoing Medically Assisted Benzodiazepine Withdrawal
Brief Title: Abuse Liability of Pregabalin and Its Effects on Benzodiazepine Withdrawal Symptoms
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low enrollment.
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Beth Sproule, Clinician Scientist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 079-2014
Record Dates: First submitted 2015-04-15; First posted 2015-04-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Substance-Related Disorders
MeSH Terms: conditions — Substance-Related Disorders | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Active Comparator): Pregabalin titrated up to, and tapered from, 225mg/day in divided doses for 10 days
  Interventions: Drug: Pregabalin; Drug: Placebo
- Placebo (Placebo Comparator): Placebo for 10 days
  Interventions: Drug: Pregabalin; Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — In replacement of their morning 75mg pregabalin or placebo dose on Days 6 and 8, all participants will receive either a single dose of 300mg of pregabalin or placebo, in a randomized, double-blind, crossover manner. This is when steady state concentrations of pregabalin occur.
  Other Names: Lyrica
Drug: Placebo — In replacement of their morning 75mg pregabalin or placebo dose on Days 6 and 8, all participants will receive either a single dose of 300mg of pregabalin or placebo, in a randomized, double-blind, crossover manner. This is when steady state concentrations of pregabalin occur.

SUMMARY:
The purpose of this study is to determine if a single dose of pregabalin 300mg in patients receiving medications for sedative-hypnotic withdrawal symptoms will produce meaningful differences in measures of "drug liking" and "drug high" as compared to placebo.

DETAILED DESCRIPTION:
Pregabalin is currently being explored as a pharmacotherapy for substance use disorders. Open-labeled, uncontrolled studies indicate modest efficacy of pregabalin in benzodiazepine withdrawal symptom management and as a long-term benzodiazepine dependence treatment. Concurrently, there is increasing information from case reports and adverse drug event registries regarding pregabalin abuse in patients with substance use disorders.

Given that the abuse liability of pregabalin has not been clearly established, nor its effects on benzodiazepine withdrawal symptoms in inpatients, this study is a randomized, double-blind, placebo-controlled, cross-over, abuse liability study of a single dose of pregabalin 300mg, nested within a randomized,double-blind placebo-controlled, feasibility study evaluating pregabalin's effects on withdrawal symptoms in inpatients undergoing medically-assisted withdrawal from benzodiazepine, zopiclone or zolpidem.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Medical Withdrawal Unit at the Centre for Addiction and Mental Health for medically assisted withdrawal from benzodiazepines, zopiclone and/or zolpidem
* Willing and capable to give written informed consent

Exclusion Criteria:

* Patients who are hypersensitive to pregabalin or to any ingredient in the formulation or component of the container.
* Pregnant or nursing women
* Renal impairment (creatinine clearance less than 60ml/min)
* History of angioedema, or taking drugs associated with angioedema (e.g., ACE-inhibitors).
* Currently taking pregabalin or gabapentin
* Currently taking thiazolidinedione antidiabetic agents (e.g., rosiglitazone, pioglitazone)
* Previous history of pregabalin or gabapentin abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline on Visual Analogue Scale for "Drug Liking" over 5 hours post-dose administration | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose

SECONDARY OUTCOMES:
Profile of Mood States (POMS) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Psychomotor Performance (Digit Symbol Substitution Test (DSST) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Digit Symbol Substitution Test (DSST)
Visual Analogue Scale for "Take Drug Again" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Any Drug Effects" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Good Effects" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Bad Effects" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Feel Sick" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Nausea" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Sleepy" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Visual Analogue Scale for "Dizzy" | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
Sedation (Addiction Research Center Inventory (ARCI) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Addiction Research Center Inventory (ARCI)
Euphoria (Addiction Research Center Inventory (ARCI) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Addiction Research Center Inventory (ARCI)
Dysphoric Changes (Addiction Research Center Inventory (ARCI) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Addiction Research Center Inventory (ARCI)
Psychotomimetic Changes (Addiction Research Center Inventory (ARCI) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Addiction Research Center Inventory (ARCI)
Somatic Disturbances (Addiction Research Center Inventory (ARCI) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Addiction Research Center Inventory (ARCI)
Sensory Disturbances (Addiction Research Center Inventory (ARCI) | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Addiction Research Center Inventory (ARCI)
Tmax Estimated peak plasma pregabalin concentration | On Days 6 and 8 only: obtained 1 hour post-dose
  Estimated peak plasma pregabalin concentration
Change from baseline on Visual Analogue Scale for "Drug High" over 5 hours | On Days 6 and 8 only: Baseline (0), and at 1, 2, 2.5, 3, 4, 5 hours post-dose
  Additional Primary Outcome

OTHER OUTCOMES:
Change in score on the Benzodiazepine Withdrawal Symptom Questionnaire | Day 0, then twice daily on Days 1 to 10 (i.e., directly before 8am dose and 3pm)
Change in score on the six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI) | Day 0, then twice daily on Days 1 to 10 (i.e., directly before 8am dose and 3pm)
Clinical Global Impression Scale - Severity | Day 0
Clinical Global Impression Scale - Improvement | Day 10
Benzodiazepine use post-discharge | 30 days post-discharge
  Assess benzodiazepine use since discharge
Pregabalin use post-discharge | 30 days post-discharge
  Assess pregabalin use since discharge

CONTACTS AND LOCATIONS:
Overall Officials: Beth Sproule, PharmD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The Centre for Addiction and Mental Health (CAMH) is the leading mental health and addictions research facility in Canada, and one of the largest in the world. — http://www.camh.ca/en/research/Pages/research.aspx